CLINICAL TRIAL: NCT05531591
Title: RCT of Neurocognitive and Neuroimaging Biomarkers: Predicting Progression Towards Dementia in Patients With Treatment-resistant Late-life Depression (OPTIMUM-Neuro RCT)
Brief Title: RCT of Brain Longitudinal Biomarker Study (OPT-Neuro RCT)
Acronym: ONR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 080-2017, 086-2016 RCT; R01MH114970 (NIH); R01MH114980 (NIH); R01MH114981 (NIH); R01MH114966-01 (NIH)
Record Dates: First submitted 2022-08-19; First posted 2022-09-08 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Depression; Dementia; Mild Cognitive Impairment; Treatment Resistant Depression; Major Depressive Disorder; Treatment-Refractory Depression; Late Life Depression; Geriatric Depression
Keywords: Comparative Effectiveness Research; Pragmatic Clinical Trials; Patient-Centered Outcomes Research; Research Clinical Trial; RCT
MeSH Terms: conditions — Depression; Dementia; Cognitive Dysfunction; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Aripiprazole; Bupropion; Lithium Carbonate; Nortriptyline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Aripiprazole Augmentation (Experimental): Augment current antidepressant treatment with aripiprazole (tablets), titrated from 2-15 mg daily based on symptom severity and side effects.
  Interventions: Drug: Aripiprazole Augmentation
- Bupropion Augmentation (Experimental): Augment current antidepressant treatment with bupropion once-daily extended release, titrated from 150-300 mg daily based on symptom severity and side effects.
  Interventions: Drug: Bupropion Augmentation
- Switch to Bupropion (Experimental): Taper from current antidepressant therapy. Start bupropion once-daily extended, titrated from 150-300 mg daily based on symptom severity and side effects.
  Interventions: Drug: Switch to bupropion
- Lithium Augmentation (Experimental): Augment current antidepressant treatment with lithium carbonate tablets starting at 300 mg daily, titrated per blood level to 0.4-0.6 mEq/L (milliequivalents/liter).
  Interventions: Drug: Lithium Augmentation
- Switch to Nortriptyline (Experimental): Taper from current antidepressant therapy. Start on nortriptyline tablets starting at 1 mg per kg of body weight daily, titrated per blood level to 80-120 ng/ml.
  Interventions: Drug: Switch to nortriptyline

INTERVENTIONS:
Drug: Aripiprazole Augmentation — Augment current antidepressant treatment with aripiprazole (tablets). Start at 2 mg daily; increase every two weeks (i.e., to 5, 7, 10 mg) to a maximum of 15 mg daily based on symptom severity and side effects.
  Other Names: Abilify
  Arms: Aripiprazole Augmentation
Drug: Bupropion Augmentation — Augment current antidepressant treatment with bupropion once-daily extended release, starting at 150 mg daily; titrated after four weeks to 300 mg daily based on symptom severity and side effects.
  Other Names: Wellbutrin
  Arms: Bupropion Augmentation
Drug: Switch to bupropion — Taper from current antidepressant therapy. Start bupropion once-daily extended release at 150 mg daily; titrated after four weeks to 300 mg daily based on symptom severity and side effects.
  Other Names: Wellbutrin
  Arms: Switch to Bupropion
Drug: Lithium Augmentation — Augment current antidepressant treatment with lithium carbonate tablets starting at 300 mg daily, titrated per blood level to 0.4-0.6 meQ/L.
  Other Names: Lithium carbonate; Eskalith
  Arms: Lithium Augmentation
Drug: Switch to nortriptyline — Taper from current antidepressant therapy. Start on nortriptyline tablets starting at 1 mg per kg of body weight daily, titrated per blood level to 80-120 ng/ml
  Other Names: Pamelor
  Arms: Switch to Nortriptyline

SUMMARY:
The purpose of this study is to assess which antidepressants work the best in older adults who have treatment-resistant depression (TRD), and to test whether treatment-resistant late life depression is associated with declines in memory and attention and brain structure and function.

DETAILED DESCRIPTION:
Older adult participants with treatment-resistant depression will be randomly assigned to a Step 1 medication strategy.

* Adding aripiprazole to current antidepressant medication
* Adding bupropion to current antideprssant medication
* Replacing current antidepressant medication with bupropion

If depression is not relieved at the end of 10 weeks, or if participants do not qualify for Step 1, participants will be randomly assigned to a Step 2 medication strategy:

* Adding lithium to current antidepressant medication
* Replacing current antidepressant medication with nortriptyline

All medication strategies will be offered in collaboration with participants' own physicians with the the research team providing support and guidance.

After treatment in Step 1 and/or Step 2, participants will enter the Continuation Phase to assess long term follow-up outcomes for 12 months.

Participants in the Optimizing Outcomes of Treatment-Resistant Depression in Older Adults (OPTIMUM) (NCT02960763) study, will also be asked to participate in this clinical trial to gather imaging and biomarker data. The study will test if changes in brain structure and function are associated with decreases in memory. In this study, investigators will conduct a series of assessments/tests, mainly brain imaging and assessments of participant's memory and attention, to better understand how depression is linked to memory and thinking in older persons.

* Investigators will be collecting blood biomarkers as part of their study procedures. These samples will be used to look at other factors that may relate to depression or memory and attention processes.
* Mechanisms of Late life depression (LLD)-dementia through functional Magnetic Resonance Imaging (fMRI): Analyzing mechanisms of the LLD-dementia relationship through fMRI acquisitions and analyses, to capture the specific brain networks implicated in executive function and episodic memory decline.
* Neuropsychological Data: Including Montreal Cognitive Assessment (MoCA), Wide Range Achievement Test-4 (WRAT-4) Reading subtest, Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) and Delis-Kaplan Executive Function System (D-KEFS) (Color Word Interference, Trail Making and Verbal Fluency).
* Clinical Scales: Including the Everyday Cognition Scale (E-Cog), Global Clinical Dementia Rating (CDR), Performance Assessment of Selfcare Skills (PASS)-Cognitive Instrumental Activities of Daily Living(CIADL) Short version, Patient Health Questionnaire (PHQ-9), and Suicide Risk Assessments (Suicide Questions, Baseline Suicidal Ideation, Suicide Intent Scale, Beck Lethality Scale, Decision Outcome Inventory, Columbia-Suicide Severity Rating Scale, and High Suicide Risk Protocol).

Investigators hope that this study will help the scientific community to understand why some people with depressive symptoms that are resistant to treatment in late-life experience declines in their memory and attention and whether effective treatment of such depression reduces that risk. Finally, investigators hope that this study will eventually lead to the development of better treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60 and older, with approximately equal proportions aged 60-70 and 70+.
* Current Major Depressive Disorder (MDD), single or recurrent, as diagnosed by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
* Failure to respond adequately to two or more antidepressant treatment trials of recommended dose and length (approximately 12 weeks).
* PHQ-9 score of 10 or higher.

Exclusion Criteria:

* Dementia; patients screened out due to possible dementia will be referred to a local Memory Clinic or back to their clinician for evaluation to clarify the presence or absence of dementia.
* Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms.
* High risk for suicide (e.g. active Suicidal ideations (SI) and or current/recent intent or plan)). Urgent psychiatric referral will be made in these cases.
* Non-correctable, clinically significant sensory impairment (e.g., cannot hear well enough to cooperate with interview).
* Unstable medical illness, including delirium, uncontrolled diabetes mellitus, hypertension, hyperlipidemia, or cerebrovascular or cardiovascular risk factors that are not under medical management.
* Moderate to severe substance or alcohol use disorder, as determined by study physician.
* Seizure disorder.
* Parkinson's Disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Well-Being | Step 1 (10 weeks), Step 2 (10 weeks), a period of up to 20 weeks
  Psychological well-being was assessed using the NIH Toolbox Psychological Wellbeing subscales of Positive Affect and General Life Satisfaction, with a T score calculated as the average of these two subscales. Higher scores indicate greater positive affect and life satisfaction. Reference T-score (mean=50, Standard Deviation (SD)=10.
Assessing the change in the Number of Participants With Remission From Depression | Step 1 (10 weeks), Step 2 (10 weeks), a period of up to 20 weeks
  Remission defined as Montgomery Asberg Depression Rating Scale score ≤10. Scale ranges from 0-60 with higher scores indicating higher depressive symptoms.
Safety Outcomes Assessment for Serious Adverse Events | Step 1 (10 weeks), Step 2 (10 weeks), a period of up to 20 weeks
  Assessing; Life threatening illness, hospitalization, or need of medical care over the duration of the study
To observe whether persistent (non-remitting) depression leads to greater cognitive decline (focusing on executive and episodic memory (EEM)-related cognitive domains | Baseline, 6-months, 24-months
  Using baseline differences to compare if non-remitters demonstrate greater decline in EEM than remitters leading to greater cognitive decline using . Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).

OTHER OUTCOMES:
Plasma biomarkers will be analyzed using a customized multiplex protein array platform for the Senescence-Associated Secretory Phenotype (SASP). | Baseline, 6-months, 24-months
  The SASP index will be used to look at circulating proteins related to immune-inflammatory control

CONTACTS AND LOCATIONS:
Overall Officials: Aristotle Voineskos, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (4):
- United States (3):
  - UCLA Late-Life Mood, Stress, and Wellness Research Program, Los Angeles, California
  - Washington University School of Medicine Healthy Mind Lab, St Louis, Missouri
  - Columbia University Adult and Late Life Depression Clinic, New York, New York
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
A cleaned, complete, and de-identified copy of the final data set including administrative and technical metadata records will be made available on the National Institute of Mental Health (NIMH) Data Archive and registered at clinicaltrials.gov.
Time Frame: Data will become available after all analyses and initial publication is complete.
Access Criteria: The data will be accessible through the NIMH Data Archive (Collection ID: 2851). Please contact the principal investigators if you have further queries about access criteria.